CLINICAL TRIAL: NCT00741702
Title: Diabetes Risk Evaluation and Microalbuminuria in Saskatchewan First Nations Peoples
Acronym: DREAM3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Pfizer (Industry)
Responsible Party: Principal Investigator, Sheldon Tobe, Principal Investigator, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 231-2001
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Hypertension; Diabetes Mellitus
Keywords: Hypertension; Type 2 diabetes; First Nations populations
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): A home care nurse followed a predefined treatment algorithm of pharmacologic antihypertensive therapy.
  Interventions: Other: Nurse administered treatment algorithm
- Control group (No Intervention): Treatment decisions were made by each subject's primary care physician. Participants in this group received usual care.

INTERVENTIONS:
Other: Nurse administered treatment algorithm — Start with Irbesartan 150 mg/d; check BP in 6 wks, if BP >=130/80 mm HF, 300 mg/d irbesartan; check BP at next visit, if BP>= 130/80 mm Hg, add HCTZ 12.5 mg/d; check BP at next visit, if BP>=130/80 mm Hg, add verapamil 180 mg/d; check BP at next visit, if BP>=13/80 mm Hg, increase verapamil to 240 mg/d
  Arms: Intervention group

SUMMARY:
This randomized controlled trial was designed to assess whether a community-based treatment strategy implemented by home care nurses would be effective in controlling hypertension in First Nations people with existing hypertension and type 2 diabetes.

DETAILED DESCRIPTION:
Two community-based strategies for controlling hypertension in First Nations people with existing hypertension and diabetes were compared. In the intervention group, a home care nurse followed a predefined treatment algorithm of pharmacologic antihypertensive therapy. In the control group, treatment decisions were made by each subject's primary care physician. The primary outcome measure was the difference between the 2 groups in teh change in systolic blood pressure after 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age>= 18 yr
* Type 2 diabetes mellitus
* Persistent hypertension (systolic pressure >= 130 mmHg, diastolic pressure >= 80 mm Hg, or both)

Exclusion Criteria:

* use of beta blocker
* women of child-bearing age not able to use a reliable method of birth control
* Connective tissue disorder
* Severe systemic or malignant disease
* Inability to follow the protocol
* Bilateral renal artery stenosis and other causes of secondary hypertension
* Serum creatinine level > 250 micromol/L
* cerebrovascular even within 6 mo
* valvular heart disease
* unstable angina
* Myocardial infarction
* Revascularization procedure within 3 mo before study recruitment
* heart failure
* cardiac arrhythmia requiring medical treatment or heart block
* active hepatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2001-09; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
systolic blood pressure | 12 months

SECONDARY OUTCOMES:
Change in diastolic blood pressure, change in urine albumin status and incidence of adverse events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Tobe, MD, FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre